CLINICAL TRIAL: NCT03164226
Title: Prognostic Value of Non-invasive Index of Endothelial Function in Emergency Department Patients With Undifferentiated Chest Pain
Brief Title: Prognostic Value of Non-invasive Index of Endothelial Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ENDOPAT
Record Dates: First submitted 2017-05-14; First posted 2017-05-23 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Chest Pain; Major Adverse Cardiovascular Events
Keywords: endothelial function; chest pain; major adverse cardiovascular events; Endo-PAT
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient consulting for chest Pain in ED (Other): Any patient ≥ 25 years consulting for chest pain in the emergency department from 8:00 am to 8:00 pm (for the unavailability of the endopat device during the guard).
  Interventions: Device: Digital plethysmography in stratifying the cardiovascular risk for patients consulting for chest pain

INTERVENTIONS:
Device: Digital plethysmography in stratifying the cardiovascular risk for patients consulting for chest pain — To verify the contribution of digital plethysmography in stratifying the cardiovascular risk for patients consulting for chest pain

SUMMARY:
The objective of this study is to determine the prognostic performance of endothelial function assessment, using endothelial peripheral arterial tonometry (Endo-PAT), associated to TIMI risk score, in patients consulting the emergency department for non-traumatic chest pain.

To determine the sensitivity, specificity, negative and positive predictive value of this method that was not previously used for this purpose.

DETAILED DESCRIPTION:
Chest pain is a frequent reason for consultation in the emergency room, which can be as much as 5 to 10% of consultants. Stratifying the cardiovascular risk for patients consulting for chest pain is sometimes difficult.

The endothelium plays a crucial role in maintaining the tone and vascular integrity and in particular the secretion of vasodilator and vasoconstrictor mediators. In most vascular pathologies, this equilibrium will be broken by the attenuation of the vasodilating function of the endothelium. This is called endothelial dysfunction.

Several tools for measuring endothelial function have been developed, the main characteristics of which are: noninvasive, reproducible, independent operators, predictive of the disease, safe for subjects, inexpensive and easy to use.

In this study we will be interested in digital plethysmography which has shown its effectiveness in:

* Screening for cardiovascular risk in asymptomatic subjects.
* The risk of a new cardiovascular event in the sick.
* Evaluation of the response to certain therapies.

Goal of the study :

The objective of this study is to to determine the prognostic performance of endothelial function assessment, using endothelial peripheral arterial tonometry (Endo-PAT), associated to TIMI risk score, in patients consulting the emergency department for non-traumatic chest pain.

To determine the sensitivity, specificity, negative and positive predictive value of this method that was not previously used for this purpose, hence the originality of this study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥ 25 years consulting for chest pain in the emergency department from 8:00 am to 8:00 pm (for the unavailability of the endopat device during the guard).

Exclusion Criteria:

* Chest pain of traumatic origin.
* Hemodynamic instability.
* Myocardial infarction requiring urgent revascularization.
* Parkinsonism: tremor problem.
* Refusal, communication problem.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Prognostic performance of Endo-PAT in predincting major adverse cardiovascular events | 30 days
  To determine the sensitivity, specificity, negative and positive predictive value of the Endopat associated to TIMI risk score in the the prediction of major adverse cardiovascular events in patients consulting the emergency department for chest pain

CONTACTS AND LOCATIONS:
Overall Officials: nouira semir, MD, Principal Investigator — University of Monastir
Locations (1):
- University hospital of Moastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided